CLINICAL TRIAL: NCT03620175
Title: A Phase One, Single Center, Open-Label, University of Miami Medical Center, 14 Day Study Evaluating the Safety, Cutaneous Tolerability, and Efficacy of TolaSure Topical Gel in Healthy Volunteers
Brief Title: Safety and Efficacy of Topical TolaSure on Skin Punch Biopsies in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMendics, LLC (Industry)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20180394
Record Dates: First submitted 2018-07-10; First posted 2018-08-08 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Wound Healing
Keywords: Healthy Participants; Skin; Dermal; Biopsy

STUDY DESIGN:
Intervention Model Description: Each patient receives each of the 4 treatment arms. It is closest to a single-subject design where each participant serves as their own control. The placement of treatments on each of the 4 wounds is randomized and assessed by a blinded outcomes assessor.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor is blinded to treatment groups and vehicle control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 Percent TolaSure Topical Gel (Active Comparator)
  Interventions: Drug: TolaSure Topical Gel
- 1.5 Percent TolaSure Topical Gel (Active Comparator)
  Interventions: Drug: TolaSure Topical Gel
- 0.5 Percent TolaSure Topical Gel (Active Comparator)
  Interventions: Drug: TolaSure Topical Gel
- Topical Vehicle Gel (Placebo Comparator)
  Interventions: Drug: TolaSure Topical Gel

INTERVENTIONS:
Drug: TolaSure Topical Gel — TolaSure topical gel is applied to skin punch biopsies daily over the course of 2 weeks.

SUMMARY:
TolaSure is a topical gel for the promotion of wound healing. This phase I study will assess the safety, tolerability and clinical effect of TolaSure when applied to skin wounds created by punch biopsy in healthy participants. A total of 26 healthy volunteers, males and females ages 18 years or older, will be enrolled. Subjects will monitored for safety and efficacy over the course of 2 weeks following daily topical administration of TolaSure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and Females > 18 years of age
* Health history review
* Physical exam
* Blood and urine clinical chemistries
* Pregnancy test
* Drug screen

Exclusion Criteria:

* Acute or chronic skin disorders (e.g. acne, psoriasis, dermatitis)
* Prone to keloids or hypertrophic scarring
* Topical or systemic antibiotics within 4 weeks of study enrollment
* Subjects with mental illnesses
* Diagnosed with Diabetes Type I/II
* Surgery within the previous 3 months (except for minor cosmetic or dental procedures)
* History of severe vitamin or mineral deficiency
* History of drug or alcohol abuse (as defined by the Investigator)
* Smoking/Vaping
* HIV/AIDS
* Consistently taking steroids and/or non-steroidal anti-inflammatory drugs
* Cancer diagnosis in the last year
* Currently receiving chemotherapy or radiation
* Women who are pregnant, nursing or planning a pregnancy
* Hyper- or hypo-pigmentation, or tattoos in the area where they will place the test fields
* Symptoms of a clinically significant illness in the four weeks before treatment application that may influence the outcome of the study
* Treatment with any investigational agent within one month before treatment application for this trial
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator, make the subject unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Blood and Urine Chemistries | Day 1, 2, 7 and 14.
  Absolute values and changes over time of clinical chemistries including; Absolute values and changes over time of clinical blood and urine chemistries including; Hematology and Coagulation, Coagulation, Serum Chemistry, and Urinalysis. Blood and urine analytes are measured on a per mL basis.
Cutaneous Tolerability | Day 1, 2, 7 and 14.
  Cutaneous tolerability will include an evaluation of erythema and edema following the modified Draize scoring system. Draize scores will be recorded and changes from baseline Draize scores will be monitored over the course of the time frame.
  Draize Scoring System. Erythema: 0-No Erythema, 1-Slight Erythema, 2-Well Defined Erythema, 3- Moderate or Severe Erythema, 4- Severe Erythema or slight eschar formation.
  Edema: 0- No Edema, 1- Very Slight Edema(barely perceptible), 2-Slight Edema (well defined edges), 3-Moderate Edema (raised >1mm), 4- Severe Edema (raised >1mm and extending beyond the area of exposure)

SECONDARY OUTCOMES:
Wound Closure | Day 1, 2, 7 and 14.
  Imaging of punch biopsies to monitor for healing and wound closure including measurement of changes in wound area (mm^2) over time will be assessed using digital imaging and analyzed using wound tracing techniques followed by the use of appropriate statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Karen McGuire, PhD, Study Director — BioMendics, LLC
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No